CLINICAL TRIAL: NCT01132976
Title: The Addition of a Goal-based Motivational Interview to Standardised Treatment as Usual to Reduce Dropouts From a Service for Patients With Personality Disorder: A Feasibility Study
Brief Title: The Personal Concerns Inventory Study (PCI)
Acronym: PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottinghamshire Healthcare NHS Trust (Other Government)
Collaborators: University of Nottingham (Other); Bangor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PB-PG-1207-15046
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Personality Disorders
Keywords: Personality disorders; Personal Concerns Inventory; Non completion
MeSH Terms: conditions — Personality Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal-based motivational interview (Active Comparator): Participants randomised to this group will receive the goal based motivational interview - Personal Concerns Inventory (PCI) in addition to treatment as usual.
  Interventions: Behavioral: Personal Concerns Inventory
- Treatment as usual (Other): Participants randomly allocated to this group will receive treatment as usual only, ie no specific motivational intervention.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Personal Concerns Inventory — This is a pre-treatment, goal-based motivational interview which helps to patients identify their life goals, and goal-value. The interview will last approximately 2 hours and will be carried out face to face with a therapist across one or two sessions.
  Arms: Goal-based motivational interview
Behavioral: Treatment as usual — No specific motivational interview
  Arms: Treatment as usual

SUMMARY:
Services for people with personality disorders are challenged by how to engage clients in therapy. High non-completion rates have major cost-efficiency implications, but more worrying is that drop-out may be associated with negative outcomes for clients. The investigators have developed a motivational intervention that helps people focus on their valued and attainable life goals and consider how therapy could help with goal attainment.One way to improve retention in treatment is to deliver pre-therapy motivational preparation interviews. The primary aim of our proposed research is to gather information to determine whether a randomised controlled trial of a goal-based motivational intervention is feasible in a community personality disorder treatment service.

DETAILED DESCRIPTION:
The investigators aim to work with community adults with personality disorder. Referrals to Nottinghamshire NHS Trust's community personality disorder service will be eligible for inclusion. After initial assessment for suitability for the service, patients will be randomised to receive the motivational interview plus treatment as usual or treatment as usual only. The investigators aim to recruit 100 participants over 1½ years. The comparison is between a motivational intervention called the Personal Concerns Inventory plus treatment as usual and and treatment as usual only in the client preparation phase. The feasibility measures are (1) the recruitment rate to a goal-based motivational interview plus treatment as usual or treatment as usual only, and (2) the acceptability of the intervention to clients and therapists. The investigators will also develop measures to assess the processes by which the intervention may have an effect, and assess the cost of the intervention compared with treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the Nottinghamshire Personality Disorder and Development Network
* Opted to attend group sessions within the Nottinghamshire Personality Disorder and Development Network
* Aged 18 or over.
* Proficiency in spoken English
* Capacity to provide valid informed consent

Exclusion Criteria:

* Currently enrolled in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Recruitment | 18 months
  A randomised controlled trial will be considered feasible if the recruitment rate to the project is 54% of all referrals (95% CI 54-64).
Acceptability to patients | 18 months
  80% of clients find the intervention acceptable in terms of its practicability and usefulness (95% CI 80-91)
Acceptability to staff | 18 months
  80% therapists report finding the intervention helpful (95% CI 80-100)

SECONDARY OUTCOMES:
The Treatment Engagement Rating Scale (TER; Drieschner & Boomsma, 2008) | 20 weeks after intervention
  This is a therapist rating scale with items addressing the client's participation, constructive use of sessions, opennness, efforts to change, making sacrifices, goal directedness, and reflection.
Client Service Receipt Inventory | 20 weeks after intervention
  Client self-report of receipt of services
Treatment attendance | 20 weeks after intervention
  Percentage sessions attended of sessions offered

CONTACTS AND LOCATIONS:
Overall Officials: Mary McMurran, Professor, Principal Investigator — University of Nottingham
Locations (1):
- Nottinghamshire Personality Disorder & Development Network, Mandala Centre, Nottingham, United Kingdom

REFERENCES:
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104
- [Derived] Bakari M, Munseri P, Francis J, Aris E, Moshiro C, Siyame D, Janabi M, Ngatoluwa M, Aboud S, Lyamuya E, Sandstrom E, Mhalu F. Experiences on recruitment and retention of volunteers in the first HIV vaccine trial in Dar es Salam, Tanzania - the phase I/II HIVIS 03 trial. BMC Public Health. 2013 Dec 9;13:1149. doi: 10.1186/1471-2458-13-1149. PMID 24321091
- [Derived] McMurran M, Cox WM, Whitham D, Hedges L. The addition of a goal-based motivational interview to treatment as usual to enhance engagement and reduce dropouts in a personality disorder treatment service: results of a feasibility study for a randomized controlled trial. Trials. 2013 Feb 17;14:50. doi: 10.1186/1745-6215-14-50. PMID 23414174
- [Derived] McMurran M, Cox WM, Coupe S, Whitham D, Hedges L. The addition of a goal-based motivational interview to standardised treatment as usual to reduce dropouts in a service for patients with personality disorder: a feasibility study. Trials. 2010 Oct 14;11:98. doi: 10.1186/1745-6215-11-98. PMID 20946651